CLINICAL TRIAL: NCT02089685
Title: A Phase 1/2 Clinical Trial to Study the Safety and Tolerability of MK-3475 + Pegylated Interferon Alfa-2b (PEG-IFN) and MK-3475 + Ipilimumab (IPI) in Subjects With Advanced Melanoma (MEL) and Renal Cell Carcinoma (RCC) (KEYNOTE 029)
Brief Title: Safety and Tolerability of Pembrolizumab (MK-3475) + Pegylated Interferon Alfa-2b and Pembrolizumab+ Ipilimumab in Participants With Advanced Melanoma or Renal Cell Carcinoma (MK-3475-029/KEYNOTE-29)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-029; MK-3475-029 (Other: Merck); KEYNOTE-29 (Other: Merck); 2013-004072-36 (EudraCT Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Results first posted 2022-05-18 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Renal Cell Carcinoma; Melanoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma | interventions — pembrolizumab; peginterferon alfa-2b; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pembrolizumab + PegIFN-2b (Experimental): Participants in Part 1A receive pembrolizumab intravenously (IV) 200 mg every three weeks (Q3W) + PEG-IFN at assigned dose subcutaneously (SC) once a week for up to ~2 years.
  Interventions: Biological: Pembrolizumab; Biological: PegIFN-2b
- Pembrolizumab + IPI Q3W (Experimental): Participants in Parts 1A and 1B receive pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks.
  Interventions: Biological: Pembrolizumab; Biological: Ipilimumab
- Pembrolizumab + IPI Q6W (Experimental): Participants in Part 1C receive pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 50 mg every 6 weeks (Q6W) for up to ~24 weeks.
  Interventions: Biological: Pembrolizumab; Biological: Ipilimumab
- Pembrolizumab + IPI Q12W (Experimental): Participants in Part 1C receive pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 100 mg every 12 weeks (Q12W) for up to ~48 weeks.
  Interventions: Biological: Pembrolizumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475
Biological: PegIFN-2b — Subcutaneous infusion
  Other Names: PegIntron®; Sylatron®
  Arms: Pembrolizumab + PegIFN-2b
Biological: Ipilimumab — IV infusion
  Other Names: Yervoy®
  Arms: Pembrolizumab + IPI Q12W; Pembrolizumab + IPI Q3W; Pembrolizumab + IPI Q6W

SUMMARY:
This study is being done to analyze the safety, tolerability, and efficacy of treatment for advanced melanoma (MEL) and renal cell carcinoma (RCC) using combination regimens of pembrolizumab + pegylated interferon alfa-2b (PegIFN-2b) and pembrolizumab + ipilimumab (IPI). The primary hypothesis is that these combinations will be sufficiently well-tolerated to permit continued clinical investigation.

DETAILED DESCRIPTION:
The trial is being done in three parts: Part 1A (MEL and RCC) will define the maximum tolerated dose (MTD)/maximum administered dose (MAD) for the drug combinations; a recommended Phase 2 dose (RP2D) for each combination will be identified. Part 1B (MEL-single arm expansion) will better characterize safety and efficacy and provide preliminary efficacy data for the pembrolizumab + IPI combination in participants with MEL. Part 1C (MEL) is added as the third part of the study with Amendment 3. Part 1C will evaluate safety and efficacy for different doses and dosing intervals for IPI in combination with pembrolizumab in participants with advanced MEL.

In the pembrolizumab + IPI study arms, qualified participants who receive the first course but experience disease progression after discontinuing pembrolizumab with stable disease or better, may, at the investigator's discretion, initiate a second course of pembrolizumab at the same dose and schedule for up to 17 doses (up to ~1 additional year) + IPI at the same dose and schedule for up to 4 doses (up to ~12 additional weeks). In the pembrolizumab + PEG-IFN study arms, qualified participants who receive the first course but experience disease progression after discontinuing pembrolizumab with stable disease or better may, at the investigator's discretion, initiate a second course of pembrolizumab at the same dose and schedule for up to 17 doses (up to ~1 additional year). Per protocol, response or progression during the second course will not count towards efficacy outcome measure and adverse events during the second course will not count towards safety outcome measures.

Part 2 (MEL and RCC) is a randomized portion of the trial and will evaluate preliminary efficacy of the drug combinations for advanced MEL participants. Part 2 was removed from the study with Amendment 3 of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of advanced/unresectable or metastatic MEL or RCC (Part 1A only) with predominantly clear cell elements
* Previously untreated stage III/IV advanced or metastatic MEL (Part 1C only)
* MEL subjects may be treatment naïve or may have received prior lines of therapy for metastatic disease (Parts 1A and 1B)
* RCC subjects must have received ≥1 prior line of therapy for metastatic disease (Part 1A)
* Measurable disease as defined by RECIST 1.1
* Must provide a tumor sample (archival or newly obtained biopsy) that is adequate for determination of PD (programmed cell death)-Ligand 1 status by immunohistochemistry at a central pathology laboratory prior to enrollment. Note: Adequacy of the tumor sample for PD-Ligand 1 testing is not required prior to enrollment in Part 1C
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function
* Resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (Parts 1A and 1B) and/or recovered from major surgery or radiation therapy
* Female participants of childbearing potential must be willing to use adequate contraception during the course of the study through 120 days after the last dose of study drug
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study drug

Exclusion Criteria

* Uveal or ocular MEL
* Prior therapy with an anti-programmed cell death (anti-PD)-1, anti-PD-Ligand 1, anti-PD-Ligand 2 or with an agent directed to another co-inhibitory T-cell receptor or has previously participated in a pembrolizumab clinical trial. Note: In Part 1C, participants may have received anti-PD-1 and/or anti-Cytotoxic T-lymphocyte-associated antigen 4 (anti-CTLA-4) as part of their neo/adjuvant treatment.
* Has received prior anti-cancer therapy, monoclonal antibody, chemotherapy, or an investigational agent or device within 4 weeks or 5 half-lives (whichever is longer) before first dose of trial drug or not recovered (≤ Grade 1 or at baseline) from AEs due to previously administered agents (Parts 1A and 1B)
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Known additional malignancy that is progressing or requires active treatment with the exception of early stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer or in situ breast cancer that has undergone potentially curative therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Severe hypersensitivity to any pembrolizumab excipients
* Active autoimmune disease requiring systemic treatment in the past 2 years
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Active infection requiring systemic therapy
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial from screening through 120 days after the last dose of study drug
* Prior therapy with interferon alfa (in neoadjuvant, adjuvant, or metastatic settings) (Part 1A only)
* Uncontrolled thyroid dysfunction
* Uncontrolled diabetes mellitus.
* Known history of human immunodeficiency virus (HIV)
* Known history of or is positive for Hepatitis B or Hepatitis C
* Received a live vaccine within 30 days prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Long GV, Atkinson V, Cebon JS, Jameson MB, Fitzharris BM, McNeil CM, Hill AG, Ribas A, Atkins MB, Thompson JA, Hwu WJ, Hodi FS, Menzies AM, Guminski AD, Kefford R, Kong BY, Tamjid B, Srivastava A, Lomax AJ, Islam M, Shu X, Ebbinghaus S, Ibrahim N, Carlino MS. Standard-dose pembrolizumab in combination with reduced-dose ipilimumab for patients with advanced melanoma (KEYNOTE-029): an open-label, phase 1b trial. Lancet Oncol. 2017 Sep;18(9):1202-1210. doi: 10.1016/S1470-2045(17)30428-X. Epub 2017 Jul 17. PMID 28729151
- [Result] Carlino MS, Menzies AM, Atkinson V, Cebon JS, Jameson MB, Fitzharris BM, McNeil CM, Hill AG, Ribas A, Atkins MB, Thompson JA, Hwu WJ, Hodi FS, Guminski AD, Kefford R, Wu H, Ibrahim N, Homet Moreno B, Long GV. Long-term Follow-up of Standard-Dose Pembrolizumab Plus Reduced-Dose Ipilimumab in Patients with Advanced Melanoma: KEYNOTE-029 Part 1B. Clin Cancer Res. 2020 Oct 1;26(19):5086-5091. doi: 10.1158/1078-0432.CCR-20-0177. Epub 2020 Jun 30. PMID 32605909
- [Derived] Atkins MB, Hodi FS, Thompson JA, McDermott DF, Hwu WJ, Lawrence DP, Dawson NA, Wong DJ, Bhatia S, James M, Jain L, Robey S, Shu X, Homet Moreno B, Perini RF, Choueiri TK, Ribas A. Pembrolizumab Plus Pegylated Interferon alfa-2b or Ipilimumab for Advanced Melanoma or Renal Cell Carcinoma: Dose-Finding Results from the Phase Ib KEYNOTE-029 Study. Clin Cancer Res. 2018 Apr 15;24(8):1805-1815. doi: 10.1158/1078-0432.CCR-17-3436. Epub 2018 Jan 22. PMID 29358500
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response or progression during the second course were not counted towards efficacy outcome measure and adverse events during the second course were not counted towards safety outcome measures.
  Part 2 of the study was not conducted.
Groups:
- Part 1A Pembrolizumab + IPI 1 mg/kg: Participants in Part 1A received pembrolizumab intravenously (IV) 200 mg every 3 weeks (Q3W) for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year + IPI at the same dose and schedule for up ~12 additional weeks.
- Part 1A Pembrolizumab + Pegylated Interferon Alfa-2b (PEG-IFN) 1 µg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W + PEG-IFN 1 µg/kg subcutaneously (SC) once a week for up to ~2 years. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year.
- Part 1A Pembrolizumab + PEG-IFN 2 µg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W + PEG-IFN 2 µg/kg SC once a week for up to ~2 years. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year.
- Part 1B Pembrolizumab + IPI 1 mg/kg: Participants in Part 1B received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year + IPI at the same dose and schedule for up ~12 additional weeks.
- Part 1C Pembrolizumab + IPI 50 mg: Participants in Part 1C received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 50 mg every 6 weeks (Q6W) for up to ~24 weeks. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year + IPI at the same dose and schedule for up ~12 additional weeks.
- Part 1C Pembrolizumab + IPI 100 mg: Participants in Part 1C received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 100 mg every 12 weeks (Q12W) for up to 48 weeks. Qualified participants who received the first course but continued to experience disease progression may have, at investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year + IPI at the same dose and schedule for up ~12 additional weeks.
Period: Overall Study
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + Pegylated Interferon Alfa-2b (PEG-IFN) 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab + IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Started | 23 | 14 | 3 | 153 | 51 | 51
Treated | 22 | 14 | 3 | 153 | 51 | 51
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 14 | 3 | 153 | 51 | 51
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Clinical Progression | 4 | 0 | 0 | 5 | 1 | 2
Not completed — Excluded Medication | 1 | 0 | 0 | 11 | 2 | 1
Not completed — Progressive disease | 13 | 10 | 3 | 51 | 17 | 12
Not completed — Follow up ended by sponsor | 2 | 2 | 0 | 70 | 26 | 26
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 8 | 1 | 1
Not completed — Status not recorded | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 7 | 2 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Screen failure | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1A Pembrolizumab + IPI 1 mg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year + IPI at the same dose and schedule for up ~12 additional weeks.
- Part 1A Pembrolizumab + Pegylated Interferon Alfa-2b (PEG-IFN) 1 µg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W + PEG-IFN 1 µg/kg SC once a week for up to ~2 years. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year.
- Part 1C Pembrolizumab + IPI 50 mg: Participants in Part 1C received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 50 mg Q6W for up to ~24 weeks. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year + IPI at the same dose and schedule for up ~12 additional weeks.
- Part 1C Pembrolizumab + IPI 100 mg: Participants in Part 1C received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 100 mg Q12W for up to 48 weeks. Qualified participants who received the first course but continued to experience disease progression may have, at investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year + IPI at the same dose and schedule for up ~12 additional weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + Pegylated Interferon Alfa-2b (PEG-IFN) 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab + IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg | Total
Number analyzed (Participants) | 23 | 14 | 3 | 153 | 51 | 51 | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (12.3) | 60.3 (10.4) | 61.7 (18.5) | 59.9 (12.5) | 60.8 (12.9) | 62.8 (11) | 60.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 0 | 52 | 13 | 18 | 98
  Male | 13 | 9 | 3 | 101 | 38 | 33 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 21 | 9 | 2 | 142 | 41 | 45 | 260
  Unknown or Not Reported | 1 | 5 | 1 | 10 | 8 | 6 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 1 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 0 | 2
  White | 19 | 13 | 1 | 150 | 42 | 46 | 271
  More than one race | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 8 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose-limiting Toxicities (DLTs) (Part 1A)
Description: Participants in Part 1A were analyzed for DLTs. DLTs included all adverse experiences that were clearly not related to disease progression or intercurrent illness if judged by the investigator to be possibly, probably, or definitely related to study intervention. Reported adverse experiences used the Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.0. DLTs were analyzed and reported separately for protocol specified clinical indications of metastatic melanoma (MEL) and renal cell carcinoma (RCC) in Part 1A: Part 1A Pembrolizumab + IPI 1mg/kg (MEL), Part 1A Pembrolizumab + IPI 1 mg/kg (RCC), Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (MEL), Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (RCC), Part 1A Pembrolizumab + PEG-IFN 2 µg/kg (RCC). Per protocol, DLT outcome analysis did not include Parts 1B and 1C.
Time Frame: Up to ~6 Weeks
Population: Participants in Part 1A with MEL and RCC who completed the first cycle of study treatment or discontinued from trial due to drug-related adverse event (DRAE). DLTs were analyzed and reported separately for protocol specified clinical indications of MEL and RCC in Part 1A. Per protocol, Parts 1B and 1C were excluded from DLT outcome analysis.
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Groups:
- Part 1A Pembrolizumab + IPI 1 mg/kg (MEL): Participants in Part 1A with MEL received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks.
- Part 1A Pembrolizumab + IPI 1 mg/kg (RCC): Participants in Part 1A with RCC received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks.
- Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (MEL): Participants in Part 1A with MEL received pembrolizumab IV 200 mg Q3W + PEG-IFN 1 µg/kg SC once a week for up to ~2 years.
- Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (RCC): Participants in Part 1A with RCC received pembrolizumab IV 200 mg Q3W + PEG-IFN 1 µg/kg SC once a week for up to ~2 years.
- Part 1A Pembrolizumab + PEG-IFN 2 µg/kg (RCC): Participants in Part 1A with RCC received pembrolizumab IV 200 mg Q3W + PEG-IFN 2 µg/kg SC once a week for up to ~2 years.
- Part 1B Pembrolizumab+ IPI 1 mg/kg: Participants in Part 1B received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks.
- Part 1C Pembrolizumab + IPI 50 mg: Participants in Part 1C received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 50 mg Q6W for up to ~24 weeks.
- Part 1C Pembrolizumab + IPI 100 mg: Participants in Part 1C received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 100 mg Q12W for up to ~48 weeks.
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg (MEL) | Part 1A Pembrolizumab + IPI 1 mg/kg (RCC) | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (MEL) | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (RCC) | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg (RCC) | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 11 | 8 | 5 | 9 | 3 | 0 | 0 | 0
Percentage of Participants | 36.4 [20.6 to 54.5] | 25 [10.2 to 45.4] | 20 [5.1 to 44.8] | 0.0 [0.0 to 14.9] | 66.7 [36.5 to 89.4] |  |  |

2. Primary Outcome: Percentage of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Reported adverse experiences used the Common Terminology for Adverse Events (CTCAE) Version 4.0.The number of participants who experienced at least one AE was reported.
Time Frame: Up to ~84 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 1A Pembrolizumab + IPI 1 mg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks.
- Part 1A Pembrolizumab + PEG-IFN 1 µg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W + PEG-IFN 1 µg/kg SC once a week for up to ~2 years.
- Part 1A Pembrolizumab + PEG-IFN 2 µg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W + PEG-IFN 2 µg/kg SC once a week for up to ~2 years.
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 22 | 14 | 3 | 153 | 51 | 51
Percentage of Participants | 100.0 | 100.0 | 100.0 | 99.3 | 100.0 | 100.0

3. Primary Outcome: Percentage of Participants Discontinuing Study Drug Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Reported adverse experiences used the CTCAE Version 4.0. The percentage of participants who discontinued study treatment due to an AE was reported.
Time Frame: Up to ~24 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 22 | 14 | 3 | 153 | 51 | 51
Percentage of Participants | 40.9 | 50.0 | 66.7 | 37.3 | 19.6 | 37.3

4. Primary Outcome: Percentage of Participants Experiencing Adverse Events of Special Interest (AEOSIs) (Parts 1B and 1C)
Description: AEOSIs consist of immune-mediated events, infusion reactions and depression. Events include Pneumonitis, Colitis, Hepatitis, Nephritis, Adrenal Insufficiency, Hypophysitis, Hyperthyroidism, Hypothyroidism, Thyroiditis, Type 1 Diabetes Mellitus, Skin Disorders, Uveitis, Pancreatitis, Myositis, Guillain-Barre Syndrome, Myocarditis, Encephalitis, Sarcoidosis, Infusion Reactions, Myasthenic Syndrome, Myelitis, Vasculitis, and Cholangitis Sclerosing. Per protocol Part 1B and Part 1C are reported. Part 1A was not included in the AEOIs outcome analysis, per protocol.
Time Frame: Up to ~84 months
Population: All randomized participants in Part 1B and Part 1C who received at least one dose of study treatment. Part 1A was not included in the AEOIs outcome analysis, per protocol.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 153 | 51 | 51
Percentage of Participants |  |  |  | 60.8 | 45.1 | 56.9

5. Primary Outcome: Percentage of Participants Experiencing Grade 3-5 Drug-related AEs (Part 1C)
Description: Participants in Part 1C who experienced grade 3-5 drug-related AEs (DRAEs) using CTCAE Version 4.0 are presented. Grade 3-5 DRAEs for Parts 1A and 1B was a secondary outcome analysis, per protocol and reported later in the record.
Time Frame: Up to ~84 months
Population: All randomized participants in Part 1C who received at least one dose of study treatment. Grade 3-5 DRAEs in Parts 1A and 1B were reported separately as a secondary outcome analysis, per protocol.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 1A Pembrolizumab + IPI 1mg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks.
Arm/Group | Part 1A Pembrolizumab + IPI 1mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 51 | 51
Percentage of Participants |  |  |  |  | 27.5 | 43.1

6. Primary Outcome: Objective Response Rate (ORR) (Part 1C)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The percentage of participants who experienced a CR or PR is presented. Per protocol, ORR in Part 1C was planned and conducted as a pre-specified primary outcome analysis. ORR in Part 1B was planned and conducted as a protocol-specified secondary outcome analysis and has been reported later in the record. Outcome analysis of ORR in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: Participants in Part 1C with measurable disease at baseline based on central independent review, who had ORR data available. Per protocol, ORR in Part 1C was planned and conducted as a pre-specified primary outcome analysis. ORR in Part 1B was planned and conducted as a protocol-specified secondary outcome analysis and has been reported later in the record. Outcome analysis of ORR in Part 1A was not planned or conducted in this study, per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 46 | 43
Percentage of Participants |  |  |  |  | 69.6 [54.2 to 82.3] | 76.7 [61.4 to 88.2]

7. Primary Outcome: Progression-free Survival (PFS) (Part 2)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS was to be assessed by independent central review per RECIST 1.1. Part 2 of the study was not conducted, based on protocol specified criteria and this Part 2 specific outcome measure could not be reported.
Time Frame: Up to ~84 months
Population: Part 2 of the study was not conducted, based on protocol specified criteria and this Part 2 specific outcome measure could not be reported.
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Objective Response Rate (ORR) (Part 1B)
Description: ORR was defined as the percentage of participants who had a CR: Disappearance of all target lesions or a PR: At least a 30% decrease in the sum of diameters of target lesions as assessed using RECIST 1.1. The percentage of participants who experienced a CR or PR is presented. Per protocol, ORR in Part 1B was planned and conducted as a pre-specified secondary outcome analysis. ORR in Part 1C was planned and conducted as a protocol-specified primary outcome analysis and has been reported earlier in the record. Outcome analysis of ORR in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: Participants in Part 1B with measurable disease at baseline based on central independent review, who had ORR data available. Per protocol, ORR in Part 1B was planned and conducted as a pre-specified secondary outcome analysis. ORR in Part 1C was planned and conducted as a protocol-specified primary outcome analysis and has been reported earlier in the record. Outcome analysis of ORR in Part 1A was not planned or conducted in this study, per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 146 | 0 | 0
Percentage of Participants |  |  |  | 65.8 [57.5 to 73.4] |  |

9. Secondary Outcome: ORR by Programmed-death Receptor-ligand 1 (PD-L1) Status Using RECIST 1.1 (Parts 1B and 1C)
Description: ORR was defined as the percentage of participants who had a CR: Disappearance of all target lesions or a PR: At least a 30% decrease in the sum of diameters of target lesions as assessed using RECIST 1.1. The percentage of participants that experienced a CR or PR by PD-L1 status is presented. PD-L1 positivity was defined as ≥1% staining in tumor and inflammatory cells, while PD-L1 negativity is defined as <1% staining. ORR for participants in Parts 1B and 1C with measurable disease at baseline based on central independent review, who had ORR data available for PD-L1+ and PD-L1- participants are presented. Outcome analysis of ORR in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: Participants in Parts 1B and 1C with measurable disease at baseline based on central independent review, who had ORR data available for PD-L1+ and PD-L1- participants. Outcome analysis of ORR in Part 1A was not planned or conducted in this study, per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 144 | 41 | 38
Percentage of Participants
  PD-L1 Positive: number analyzed (Participants) | 0 | 0 | 0 | 121 | 28 | 27
  PD-L1 Positive |  |  |  | 67.8 [58.7 to 76.0] | 75.0 [55.1 to 89.3] | 85.2 [66.3 to 95.8]
  PD-L1 Negative: number analyzed (Participants) | 0 | 0 | 0 | 23 | 13 | 11
  PD-L1 Negative |  |  |  | 52.2 [30.6 to 73.2] | 53.8 [25.1 to 80.8] | 63.6 [30.8 to 89.1]

10. Secondary Outcome: Percentage of Participants With an Ordinal Response, Estimated by a Best Overall Response of VGPR or MPR (Parts 1B and 1C)
Description: Ordinal response, per RECIST 1.1 included the best overall responses of Very Good Partial Response ([VGPR]>60% tumor reduction) as well as Moderate Partial Response ([MPR]>30%- ≤60% tumor reduction). The percentage of participants in Part 1B and 1C who experienced a MPR or VGPR (based on the degree of tumor shrinkage) in participants with advanced melanoma is presented. Outcome analysis of ordinal response in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: All randomized participants in Part 1B and Part 1C who received at least one dose of study treatment and had data available for VGPR or MPR. Outcome analysis of ordinal response in Part 1A was not planned or conducted in this study, per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 146 | 46 | 43
Percentage of Participants
  MPR |  |  |  | 6.2 [2.9 to 11.4] | 8.7 [2.4 to 20.8] | 23.3 [11.8 to 38.6]
  VGPR |  |  |  | 24.0 [17.3 to 31.7] | 28.3 [16.0 to 43.5] | 20.9 [10.0 to 36.0]

11. Secondary Outcome: Duration of Response (DOR) (Parts 1B and 1C)
Description: DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on central imaging review with confirmation. The DOR as assessed using RECIST 1.1 for participants with measurable disease at baseline based on central independent review in Parts 1B and 1C who experienced a confirmed CR or PR with DOR data available is presented. Outcome analysis of DOR in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: Participants in Parts 1B and 1C with measurable disease at baseline based on central independent review, who had a confirmed CR or PR, with DOR data available. Outcome analysis of DOR in Part 1A was not planned or conducted in this study, per protocol.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 96 | 32 | 33
Months |  |  |  | NA [NA to NA] — Median and range lower and upper limit not reached. No progressive disease by the time of last disease assessment. | NA [NA to NA] — Median and range lower and upper limit not reached. No progressive disease by the time of last disease assessment. | NA [3.8 to NA] — Median and range upper limit not reached. No progressive disease by the time of last disease assessment.

12. Secondary Outcome: Progression-free Survival (PFS) (Parts 1B and 1C)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS as assessed by independent central review per RECIST 1.1 for all participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had PFS data available is presented. Outcome analysis of PFS in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: All participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had PFS data available. Outcome analysis of PFS in Part 1A was not planned or conducted in this study, per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 153 | 51 | 51
Months |  |  |  | NA [36.4 to NA] — Median and range upper limit of PFS was not reached. No progressive disease by the time of last disease assessment. | NA [14.1 to NA] — Median and range upper limit of PFS was not reached. No progressive disease by the time of last disease assessment. | NA [31.9 to NA] — Median and range upper limit of PFS was not reached. No progressive disease by the time of last disease assessment.

13. Secondary Outcome: Overall Survival (OS) (Parts 1B and 1C)
Description: OS was defined as the time from randomization to death due to any cause. OS for all participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had OS data available is presented. Outcome analysis of OS in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: All participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had OS data available. Outcome analysis of OS in Part 1A was not planned or conducted in this study, per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 1B Pembrolizumab + IPI 1 mg/kg: Participants in Part 1B received pembrolizumab IV 200 mg Q3W for up to ~2 years + IPI IV 1 mg/kg Q3W for up to ~12 weeks.
Arm/Group | Part 1A Pembrolizumab + IPI 1mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab + IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 153 | 51 | 51
Months |  |  |  | NA [NA to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events. | NA [NA to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events. | NA [39.6 to NA] — Median and range upper limits not reached due to insufficient number of OS events.

14. Secondary Outcome: PFS by PD-L1 Status Using RECIST 1.1 (Parts 1B and 1C)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PD-L1 positivity was defined as ≥1% staining in tumor and inflammatory cells, while PD-L1 negativity is defined as <1% staining. PFS for all participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had PFS data available for PD-L1+ and PD-L1- participants is presented. Outcome analysis of PFS in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: All participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had PFS data available for PD-L1+ and PD-L1- participants. Outcome analysis of PFS in Part 1A was not planned or conducted in this study, per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab + IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 151 | 46 | 44
Months
  PD-L1 Positive: number analyzed (Participants) | 0 | 0 | 0 | 127 | 32 | 31
  PD-L1 Positive |  |  |  | NA [41.6 to NA] — Median and range upper limit not reached. No progressive disease by the time of last disease assessment. | NA [NA to NA] — Median and range lower and upper limit not reached. No progressive disease by the time of last disease assessment. | NA [35.7 to NA] — Median and range upper limit not reached. No progressive disease by the time of last disease assessment.
  PD-L1 Negative: number analyzed (Participants) | 0 | 0 | 0 | 24 | 14 | 13
  PD-L1 Negative |  |  |  | 20.7 [2.8 to NA] — Range upper limit not reached. No progressive disease by the time of last disease assessment. | 23.1 [1.4 to NA] — Range upper limit not reached. No progressive disease by the time of last disease assessment. | 13.8 [1.4 to NA] — Range upper limit not reached. No progressive disease by the time of last disease assessment.

15. Secondary Outcome: OS by PD-L1 Status Using RECIST 1.1 (Parts 1B and 1C)
Description: OS was defined as the time from randomization to death due to any cause. PD-L1 positivity was defined as ≥1% staining in tumor and inflammatory cells, while PD-L1 negativity is defined as <1% staining. OS for all participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had OS data available for PD-L1+ and PD-L1- participants is presented. Outcome analysis of OS in Part 1A was not planned or conducted in this study, per protocol.
Time Frame: Up to ~84 months
Population: All participants who received at least one dose of study treatment in Part 1B and all randomized participants in Part 1C, who had OS data available for PD-L1+ and PD-L1- participants. Outcome analysis of OS in Part 1A was not planned or conducted in this study, per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab + IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 151 | 46 | 44
Months
  PD-L1 Positive: number analyzed (Participants) | 0 | 0 | 0 | 127 | 32 | 31
  PD-L1 Positive |  |  |  | NA [NA to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events. | NA [NA to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events. | NA [NA to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events.
  PD-L1 Negative: number analyzed (Participants) | 0 | 0 | 0 | 24 | 14 | 13
  PD-L1 Negative |  |  |  | NA [14.1 to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events. | 32.8 [12.9 to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events. | NA [7.6 to NA] — Median and range lower and upper limits not reached due to insufficient number of OS events.

16. Secondary Outcome: Percentage of Participants Experiencing Grade 3-5 DRAEs (Parts 1A and 1B)
Description: Participants in Parts 1A and 1B who experienced DRAEs using CTCAE Version 4.0 are presented. Grade 3-5 DRAEs for Part 1C was a primary outcome analysis, per protocol and reported earlier in the record.
Time Frame: Up to ~84 months
Population: All randomized participants in Parts 1A and 1B who received at least one dose of study treatment. Grade 3-5 DRAEs in Part 1C were reported separately as a primary outcome analysis, per protocol.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab + IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 22 | 14 | 3 | 153 | 0 | 0
Percentage of Participants | 90.9 | 71.4 | 66.7 | 70.6 |  |

17. Secondary Outcome: ORR (Part 2)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. Part 2 of the study was not conducted, based on protocol specified criteria and this Part 2 specific outcome measure was not reported.
Time Frame: Up to ~84 months
Population: as for outcome 7
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab+ IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 84 months (through database cutoff date of 01-April-2021).
Description: All-cause mortality: All randomized participants. Safety: All randomized participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Part 1A Pembrolizumab + PEG-IFN 1 µg/kg: Participants in Part 1A received pembrolizumab IV 200 mg Q3W + PEG-IFN 1 µg/kg SC once a week for up to ~2 years. Qualified participants who received the first course but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year.
Arm/Group | Part 1A Pembrolizumab + IPI 1 mg/kg | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg | Part 1B Pembrolizumab + IPI 1 mg/kg | Part 1C Pembrolizumab + IPI 50 mg | Part 1C Pembrolizumab + IPI 100 mg
All-Cause Mortality (participants affected / at risk) | 16/23 | 10/14 | 2/3 | 51/153 | 14/51 | 17/51
Serious Adverse Events (participants affected / at risk) | 9/22 | 9/14 | 2/3 | 78/153 | 26/51 | 25/51
Other Adverse Events (participants affected / at risk) | 22/22 | 14/14 | 3/3 | 152/153 | 51/51 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Pembrolizumab + IPI 1 mg/kg (N=22) | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (N=14) | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg (N=3) | Part 1B Pembrolizumab + IPI 1 mg/kg (N=153) | Part 1C Pembrolizumab + IPI 50 mg (N=51) | Part 1C Pembrolizumab + IPI 100 mg (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrotising scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic vascular thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (3)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Auditory nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
IIIrd nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Pembrolizumab + IPI 1 mg/kg (N=22) | Part 1A Pembrolizumab + PEG-IFN 1 µg/kg (N=14) | Part 1A Pembrolizumab + PEG-IFN 2 µg/kg (N=3) | Part 1B Pembrolizumab + IPI 1 mg/kg (N=153) | Part 1C Pembrolizumab + IPI 50 mg (N=51) | Part 1C Pembrolizumab + IPI 100 mg (N=51)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (14) | 0 (0) | 6 (10) | 2 (2) | 8 (13)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 0 (0) | 14 (14) | 4 (4) | 3 (3)
Hypophysitis (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0) | 13 (13) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0) | 27 (28) | 8 (9) | 10 (10)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (7) | 5 (5) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 10 (12) | 4 (4) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 6 (8) | 2 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 3 (3) | 0 (0) | 22 (25) | 7 (9) | 12 (18)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 10 (13) | 7 (9) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 4 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (3) | 0 (0) | 33 (41) | 9 (11) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 6 (12) | 5 (8) | 2 (4) | 60 (125) | 23 (41) | 24 (57)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 34 (34) | 6 (6) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 5 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 9 (13) | 2 (2) | 3 (4)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (9) | 1 (2) | 59 (78) | 14 (17) | 23 (29)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retching (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (2) | 35 (44) | 7 (8) | 12 (14)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (11) | 4 (5)
Chest pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 6 (6) | 2 (2) | 2 (3)
Chills (General disorders) | 2 (2) | 5 (9) | 2 (3) | 11 (13) | 6 (6) | 0 (0)
Fatigue (General disorders) | 9 (12) | 11 (17) | 3 (3) | 89 (117) | 31 (51) | 34 (43)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 3 (7) | 1 (1) | 23 (37) | 11 (15) | 10 (13)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (5) | 6 (7) | 5 (6)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 5 (12) | 2 (3) | 20 (25) | 7 (10) | 3 (3)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 1 (1) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (5)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 4 (4) | 5 (5)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (5) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 12 (14) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 13 (16) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 4 (6) | 3 (4)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 8 (8) | 1 (1) | 2 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 6 (7) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 17 (22) | 5 (6) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 36 (50) | 9 (10) | 8 (10)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 15 (19) | 1 (3) | 6 (7)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 3 (3) | 2 (3) | 24 (28) | 10 (19) | 6 (7)
Amylase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 30 (35) | 2 (2) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 4 (5) | 2 (3) | 20 (24) | 10 (12) | 7 (9)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 3 (5) | 0 (0) | 10 (10) | 2 (2) | 4 (8)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 3 (5) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 12 (13) | 3 (3) | 3 (3)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 3 (3) | 4 (4)
Lipase increased (Investigations) | 4 (10) | 1 (1) | 1 (1) | 39 (55) | 11 (14) | 14 (21)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 5 (13) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (8) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 6 (7) | 1 (1) | 3 (3)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 6 (7) | 1 (1) | 29 (32) | 8 (8) | 14 (14)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (10) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 2 (4) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 3 (5) | 0 (0) | 1 (1) | 1 (3) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (3) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (12) | 3 (5) | 1 (1) | 41 (58) | 19 (27) | 22 (34)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (2) | 16 (18) | 9 (9) | 8 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 1 (1) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 9 (10) | 3 (3) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 11 (11) | 5 (5) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (2) | 1 (1) | 20 (22) | 9 (16) | 9 (13)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 14 (14) | 8 (10) | 4 (4)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 3 (6) | 1 (1) | 22 (25) | 5 (5) | 5 (6)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 6 (10) | 1 (2) | 56 (68) | 15 (20) | 16 (28)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 14 (15) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 1 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 8 (9) | 1 (2) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0) | 10 (10) | 2 (2) | 4 (4)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (5) | 0 (0) | 18 (19) | 12 (16) | 10 (11)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 9 (12) | 2 (2) | 38 (47) | 17 (20) | 11 (15)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1) | 20 (26) | 9 (12) | 5 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 5 (5) | 5 (5) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 16 (17) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 16 (17) | 2 (2) | 3 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 2 (2) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 11 (11) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (3) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 7 (7) | 2 (2) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (7) | 2 (3) | 71 (98) | 19 (30) | 30 (43)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (7) | 2 (3) | 73 (120) | 27 (47) | 24 (49)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (9) | 5 (5) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 22 (28) | 3 (3) | 4 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 7 (11) | 9 (13)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (8) | 2 (2) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 31 (31) | 7 (7) | 7 (7)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 8 (8) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (2) | 0 (0) | 4 (5) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT02089685/Prot_SAP_000.pdf